CLINICAL TRIAL: NCT01550679
Title: Early Detection of COPD Patients in GOLD 0 (Smokers) Population
Acronym: MARKO
Status: Completed | Type: Observational
Sponsor: Children's Hospital Srebrnjak (Other)
Collaborators: GlaxoSmithKline (Industry); University Hospital Rijeka (Other); Clinical Hospital Center, Split (Other); General Hospital Dubrovnik (Other); Institute for Medical Research and Occupational Health, Zagreb (Unknown); Osijek University Hospital (Other)
Responsible Party: Principal Investigator, Davor Plavec, Assist.Prof., MD, PhD, Children's Hospital Srebrnjak
Other Study IDs: CHSCRT114338; GSK eTrack number CRT114338 (Other Grant/Funding Number: GlaxoSmithKline (GSK))
Record Dates: First submitted 2012-02-28; First posted 2012-03-12 (Estimated); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COPD; Smoking; Other Diagnoses, Comorbidities, and Complications
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Smokers or ex-smokers: Smokers or ex-smokers 40-65 years of age with a smoking history of at least 20 pack-years with no diagnosis of COPD or asthma

SUMMARY:
Even though the main risk factor for the development of chronic obstructive pulmonary disease (COPD) is smoking only in less than one third of the smokers the clinically manifest COPD will develop. The disease progressive nature with high disability and mortality especially in the final stages makes it plausible to detect the disease as early as possible thus allowing for the early intervention. Major intervention trials in COPD, "Towards a Revolution in COPD Health" (TORCH), "Investigating New Standards for Prophylaxis in Reducing Exacerbations" (INSPIRE), and "Understanding Potential Long-term Impacts on Function with Tiotropium" (UPLIFT) have recently shown that the beneficial impact of intervention was larger in patients being treated in earlier stages of the disease development. Till now the only tool for an early diagnosis and early intervention that could be used on the global scale was spirometry even though symptoms and deprivation of quality of life (QoL) precedes clinically relevant spirometric changes. So there is a need for a new simple tool that would allow detection of patients in a very early stage of COPD.

So the aim of this study is the development of diagnostic tools for an early detection of COPD, even before the significant change in spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Smokers or ex-smokers
* 40-65 years of age
* at least 20 pack-years of smoking history

Exclusion Criteria:

* any clinically relevant chronic disorder with a significant influence on QoL
* immuno-suppressive treatment
* significant acute respiratory disorder during last 4 weeks
* hospitalization during last 3 months
* acute myocardial information, cerebro-vascular infarction or transient ishemic attack during last 6 months
* asthma
* unable to perform the study protocol (diagnostic workout)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2010-10; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Inner consistency, repeatability, intelligibility, and applicability of MARKO questionnaire | 4 weeks after recruitment visit (2 yrs after start of recruitment)
  MARKO questionnaire will be tested for inner consistency, repeatability, intelligibility, applicability after the patient is diagnosed as having COPD and staged for severity of COPD by pulmologist. Patients will be tested twice using the same MARKO QoL questionnaire: first time at the recruitment at the primary health clinic and the second time at pulmologist office. It will be tested for it's potential to differentiate between patients with different stages of COPD.
Discriminative power of MARKO questionnaire combined with screening lung function measurement for diagnosis of COPD | 4 weeks after recruitment visit (2 yrs after start of recruitment)
  Discriminative power of MARKO questionnaire combined with screening lung function measurement using COPD6 lung function screening apparatus will be assessed for different stages of COPD based on the assessment of the diagnosis and staging of COPD made by pulmologist according to Global initiative for chronic Obstructive Lung Disease (GOLD) guidelines.
The percentage of patients progressing from GOLD 0 stage to GOLD I stage or higher | After 2 years, 3 years, and 5 years of follow-up
  The percentage of patients progressing from GOLD 0 stage to GOLD I stage or higher will be assessed based on two evaluation by pulmologist: the first one 4 weeks after recruitment when diagnosis and staging of COPD will be made and the second one after 2 (3,5) years of follow up of patient in stages GOLD 0 and I. Patients will be characterized as GOLD 0 on the first visit if they are eligible for the study and have the lung function within the normal range or as GOLD I if they have FEV1/FVC <0.7 and FEV1 >80% of normal.
Discriminative power of MARKO questionnaire combined with screening lung function measurement for an early diagnosis of COPD | After 2 years, 3 years, and 5 years of follow-up
  Discriminative power of MARKO questionnaire combined with screening lung function measurement using COPD6 lung function screening device will be assessed for an early diagnosis of COPD based on the comparison of two groups of patients: patients progressing from GOLD 0 stage to GOLD I stage or higher after 2 (3, 5) years of follow-up based on the evaluation by pulmologist according to GOLD guidelines. Patients will be characterized as GOLD 0 if they have the lung function within the normal range or as GOLD I if they have FEV1/FVC <0.7 and FEV1 >80% of normal.

SECONDARY OUTCOMES:
Prevalence of concomitant disorders in this population | 4 weeks after recruitment visit (2 yrs after start of recruitment)
Sensitivity of diagnostic parameters for early impairment in COPD | 4 weeks after recruitment visit (2 yrs after start of recruitment)
  Diagnostic parameters will be assessed after the finish of recruitment for their sensitivity for an early impairment in COPD. The sensitivity will be assessed based on their discriminative power between COPD stages 0 and I.
Predictability of developed screening questionnaire (MARKO questionnaire), and markers of early impairment in COPD for the progression of COPD | After 2 years, 3 years, and 5 years of follow-up
Comparison of MARKO questionnaire with other diagnostic tools used for evaluation of patients | After 2 years, 3 years, and 5 years of follow-up
  MARKO QoL questionnaire will be compared with other diagnostic tools used for evaluation of COPD patients (medical history, physical examination, spirometry parameters, diffusion capacity of lungs for carbon monoxide (DLCO), 6 minute walk test, The St George's Respiratory Questionnaire (SGRQ), lung function measured with COPD6 lung function screening device, COPD Assessment Test (CAT))
Prevalence of different stages of COPD (specifically GOLD stages 0 and I) in the population at risk for COPD and in general population | 4 weeks after recruitment visit (2 yrs after start of recruitment)

CONTACTS AND LOCATIONS:
Overall Officials: Davor Plavec, MD, PhD, Principal Investigator — Children's Hospital Srebrnjak; Žarko Vrbica, MD, MSc, Principal Investigator — General Hospital Dubrovnik
Locations (6):
- Croatia (6):
  - University Hospital Osijek, Osijek, Slavonsko-Baranjska
  - General Hospital Dubrovnik, Dubrovnik
  - University Hospital Rijeka, Rijeka
  - Clinical Hospital Center, Split, Split
  - Children's Hospital Srebrnjak, Zagreb
  - Institute for Medical Research and Occupational Health, Zagreb, Zagreb

REFERENCES:
- [Derived] Vrbica Z, Labor M, Gudelj I, Labor S, Juric I, Plavec D; MARKO study group. Early detection of COPD patients in GOLD 0 population: an observational non-interventional cohort study - MARKO study. BMC Pulm Med. 2017 Feb 10;17(1):36. doi: 10.1186/s12890-017-0378-6. PMID 28187733
- [Derived] Labor M, Vrbica Z, Gudelj I, Labor S, Plavec D. Diagnostic accuracy of a pocket screening spirometer in diagnosing chronic obstructive pulmonary disease in general practice: a cross sectional validation study using tertiary care as a reference. BMC Fam Pract. 2016 Aug 19;17(1):112. doi: 10.1186/s12875-016-0518-8. PMID 27542843